CLINICAL TRIAL: NCT02405156
Title: A Prospective Double-Blind, Randomized, Placebo-Controlled Trial on the Use of Letrozole Pretreatment With Misoprostol for Second-Trimester Medical Abortion
Brief Title: Letrozole Pretreatment With Misoprostol for Second-Trimester Medical Abortion
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Mohamed Samir Sweed, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 305172
Record Dates: First submitted 2015-03-16; First posted 2015-04-01 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Miscarriage
Keywords: Letrozole; misoprostol; second trimester miscarriage
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Letrozole; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- letrozole + misoprostol (Experimental): Women will receive three tablets of letrozole vaginal as a single dose, each tablet 2.5 mg (total dose 7.5 mg per day) for three days and will be followed by 200 mcg vaginal misoprostol or 100mcg vaginal misoprostol (according gestational age) soaked with saline every six hours up to maximum four doses.
  Interventions: Drug: Letrozole; Drug: Misoprostol
- placebo + misoprostol (Placebo Comparator): Women will receive three tablets of placebo vaginal as a single dose, for three days and will be followed by 200 mcg vaginal misoprostol or 100 mcg vaginal misoprostol (according gestational age) soaked with saline every six hours up to maximum four doses.
  Interventions: Drug: Placebo; Drug: Misoprostol

INTERVENTIONS:
Drug: Letrozole
  Other Names: femara
  Arms: letrozole + misoprostol
Drug: Placebo
  Arms: placebo + misoprostol
Drug: Misoprostol

SUMMARY:
To compare the success rate of letrozole and misoprostol versus misoprostol alone for medical termination of pregnancy in second trimester abortion.

DETAILED DESCRIPTION:
This prospective double-blind, randomized, clinical trial, will be conducted at Ain Shams University Maternity Hospital.

Patients fulfilling inclusion and exclusion criteria will be divided into two groups.

Group (A):

181 women will receive three tablets of letrozole (On December 28, 2005, the U.S. Food and Drug Administration approved letrozole tablets (Femara®, made by Novartis Pharmaceuticals Corp.) as a single dose, each tablet 2.5 mg (total dose 7.5 mg per day) for two days at home and will be told to bring back the empty packs. The third dose will be given on admission to hospital on day three and will be followed by 400 mcg vaginal misoprostol soaked with saline every three hours up to maximum five doses on Day 3.

Group (B):

181 women will receive three tablets of placebo (manufactured by Egyptian Group Company for drug industries) as a single dose, for two days at home and will be told to bring back the empty packs. The third dose will be given on admission to hospital on day three and will be followed by 400 mcg vaginal misoprostol soaked with saline every three hours up to maximum five doses on Day 3.

Data recording:

1. Duration of complete abortion.
2. Post abortion bleeding.
3. Incomplete delivery of the placenta necessitates evacuation under anesthesia.
4. Hemoglobin and hematocrit after 24 hours from abortion to estimate the decrease in hemoglobin level.
5. Recording maternal morbidities.
6. Patients that will receive 5 doses and did not abort till 24 hours from the first dose of misoprostol will be considered failed induction and will stop follow up without reporting outcome.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age more than 18 years old (age of legal consent).
* Gestational age between 12 weeks and 24 weeks.
* Hemoglobin >10 g/dL.
* BMI between 25 kg/m2 and 35 kg/m2.
* Miscarriage .
* Living fetus with multiple congenital malformations incompatible with life.
* PPROMs with drained liquor and parents are consenting for termination of pregnancy.

Exclusion Criteria:

* Maternal age less than 18 years old.
* Gestational age less than 12 weeks or more than 24 weeks.
* Hemoglobin <10 g/dL.
* Scared uterus (previous myomectomy, cesarean section, hysterectomy and ruptured uterus).
* Polyhydraminos.
* Anencephaly.
* Fibroid uterus.
* BMI less than 25kg/m2 and more than 35kg/m2.
* Coagulopathy.
* History or evidence of adrenal pathology.
* Previous attempts for induction of abortion in the current pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Duration of induction of abortion | 24 hours

SECONDARY OUTCOMES:
The incidence of need for surgical evacuation of placenta. | 24 hours
Hemoglobin change | 24 hours
Maternal morbidity | 24 hours
Success of induction of abortion | 24 hours
  number of participants with Success of induction of abortion
Hematocrit change | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Gomaa, MD, Principal Investigator — Ain Shams University; Ihab Serag-ElDin, MD, Study Director — Ain Shams University; Gasser El-Bishry, FRCOG, Study Director — Ain Shams University; Ahmed Swidan, M.B.B.ch, Principal Investigator — Ain Shams University; Mohamed S. Sweed, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt